CLINICAL TRIAL: NCT00954668
Title: ImmeDiate Versus EArLy Invasive Approach in Non-ST-Elevation Myocardial Infarction (IDEAL NSTEMI)
Acronym: IDEAL NSTEMI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding
Sponsor: University of Leipzig (Other)
Collaborators: Stiftung Institut fuer Herzinfarktforschung (Other)
Responsible Party: Principal Investigator, Holger Thiele, Clinical Professor Prof. Dr. Holger Thiele, University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDEAL NSTEMI 1
Record Dates: First submitted 2009-08-06; First posted 2009-08-07 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Non-ST-elevation Myocardial Infarction
Keywords: Non-ST-elevation myocardial infarction; angiography; percutaneous coronary intervention; timing
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immediate angiography (Experimental): Immediate invasive angiography < 2 h after randomization
  Interventions: Procedure: immediate angiography and revascularization
- early invasive angiography (Active Comparator): early invasive angiography 12-72 h after randomization
  Interventions: Procedure: early invasive angiography

INTERVENTIONS:
Procedure: immediate angiography and revascularization — immediate angiography < 2 hours after randomization
  Arms: immediate angiography
Procedure: early invasive angiography — early invasive angiography 12-72 h after randomization
  Arms: early invasive angiography

SUMMARY:
Of estimated 140,000 cases of acute myocardial infarction admitted to hospitals in Germany per year, approximately 50% present with Non-ST-elevation myocardial infarction (NSTEMI). The currently available evidence led to current guideline recommendations that a systematic approach of immediate angiography in NSTEMI patients stabilized with contemporary antiplatelet treatment is not mandatory. However, this immediate invasive approach is appealing because it allows treating the underlying cause (the plaque rupture) as early as possible with subsequent reduction of death and recurrent myocardial infarction. In the IDEAL NSTEMI trial we test an immediate invasive approach (<2 h) with an approach 12-72 h according top guidelines with respect to 6 months death and mortality.

ELIGIBILITY:
Inclusion Criteria:

* NSTEMI with

  * ischemic symptoms >10 minutes within 24 h
  * elevated troponin or creatine kinase above the upper limit of normal
  * ST-segment depression or transient ST-segment elevation, T-wave inversion
  * informed consent.

Exclusion Criteria:

* Age < 18 years
* Age > 90 years
* persistent angina
* hemodynamic instability
* overt congestive heart failure
* life-threatening arrhythmias
* STEMI
* limited life-expectancy < 6 months
* chronic oral anticoagulation
* fibrinolysis < 48 hours
* PCI < 14 days
* contraindication for treatment with glycoprotein IIb/IIIa inhibitors, heparin, aspirin and clopidogrel
* recent major trauma or surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2009-01-01 (Actual); Study Completion 2009-01-01 (Actual)

PRIMARY OUTCOMES:
Death and non-fatal recurrent infarction | 6 months

SECONDARY OUTCOMES:
Composite of death, recurrent non-fatal myocardial infarction, refractory ischemia or target vessel re-vascularization | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Holger Thiele, MD, Study Chair — Heart Center Leipzig - University Hospital; Uwe Zeymer, MD, Study Director — Institut für Herzinfarktforschung
Locations (1):
- University of Leipzig - Heart Center, Leipzig, Germany

IPD SHARING:
Plan to Share IPD: No